CLINICAL TRIAL: NCT04332510
Title: Acute Metabolic Effect of Different Infant Formulas (Intact Protein, Partially Hydrolyzed Protein and High Level of Partially Hydrolyzed Protein) and Breast Milk in Healthy Adults
Brief Title: A Study to Investigate the Effect of Protein in Infant Formula on Insulin Response in Adults
Acronym: IDEFIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 11.19.MET
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: To Compare the Metabolic Effects of Different Infant Milks
Keywords: infant formula; intact protein; partially-hydrolyzed protein; glucose; insulin; metabolic response
MeSH Terms: conditions — Insulin Resistance | interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: **Note: Human breast milk samples were not blinded for the care provider as they were supplied in different containers to the other milks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infant milk 1 (Experimental)
  Interventions: Other: Intact formula
- Infant milk 2 (Experimental)
  Interventions: Other: Partially hydrolyzed formula
- Infant milk 3 (Experimental)
  Interventions: Other: High protein formula
- Infant milk 4 (Experimental)
  Interventions: Other: Human breast milk

INTERVENTIONS:
Other: Intact formula — 600 ml of infant formula with intact protein
  Arms: Infant milk 1
Other: Partially hydrolyzed formula — 600 ml of infant formula with partially hydrolyzed protein
  Arms: Infant milk 2
Other: High protein formula — 600 ml of infant formula with high protein level
  Arms: Infant milk 3
Other: Human breast milk — 600 ml of breast milk, safe for human consumption
  Arms: Infant milk 4

SUMMARY:
It has been established that the consumption of a diet that causes a low rise in blood insulin levels is beneficial in terms of risk for diabetes and heart disease. Furthermore, it is known that certain nutrients contained within a food play an important role in the insulin response of that food. For example, the type and quantity of protein has been shown to affect the insulin response to particular foods.

Different types of infant formula exist, containing different levels and types of protein, yet the impact of these different infant formulas on blood insulin levels is not known.

Using a randomized, double blind, cross-over study design, the insulin response to four test milks was compared in healthy adults. The four test milks were as follows: i) infant formula containing partially hydrolyzed protein; ii) infant formula with intact protein; (iii) infant formula with a higher energy and protein content compared to (i) and (ii); and (iv) human breast milk (in a small sub-group). The aim of the study was to show that the insulin response to the partially hydrolyzed formula is similar to that of an infant formula with intact protein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 20-50 years at time of the enrollment
* Normal body weight. BMI 19-25 kg/m2
* Having obtained his/her signed informed consent

Exclusion Criteria:

Chronic or acute diseases affecting metabolism (diabetes, renal insufficiency, CVD, liver disease), dyslipidemia, as checked using the medical questionnaire and based on a biochemical blood analysis (glucose, triglycerides, cholesterol, transaminases and Gamma-GT, CRP in fasting

* Anemia (Erythrocytes < 4,6 T/l (male) or < 4,2 T/l (women); Hemoglobin Hb < 13 g/dl (male) or Hb < 12 g/dl (women); Hematocrit Ht < 40% (male) or Ht < 37% (women); sera iron < 0,6 mg/l or plasma ferritin < 120 μg /l (male) or < 60 μg/l (non menopaused women)
* Recent major surgery (3 months)
* History of cancer within the past year
* Significant weight loss during the last 3 months (more than 5% of BW)
* Regular intensive physical activity of more than 3 times of 45 min per week
* Food allergy, lactose intolerance
* Under chronic medications (except contraceptive pills) Have a regular higher alcohol consumption than 1 drink/day or occasional 1-2 drinks during week end
* Consumption of illicit drugs, as checked by a urinary testing
* Smoking (more than 5 cigarettes a day)
* Women pregnant or lactating
* Special weight reduction program /diet
* Blood donation of at least 300mL during the last 3 months or planned blood donation before the end of the study
* Subject who cannot be expected to comply with the study procedures, including consuming the test products (600 mL of milk within 10 minutes)
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Insulin response to infant formulas containing partially hydrolyzed or intact protein | 0, 15, 30, 45, 60, 90, 120, 150, 180 mins
  To show that the insulin Cmax response to a partially hydrolyzed formula is similar to that of an infant formula with intact protein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahkhalili Y, Monnard C, Grathwohl D, Sauser J, Beaumont M, Zufferey CA, Mace K. Comparison of the acute metabolic effect of different infant formulas and human milk in healthy adults: a randomized trial. Nutr Diabetes. 2021 Apr 15;11(1):13. doi: 10.1038/s41387-021-00154-3. PMID 33859173